CLINICAL TRIAL: NCT00044902
Title: Monoclonal Antibody Treatment for Non-Hodgkin's Lymphoma (Low-Grade)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Purpose: Treatment
Other Study IDs: 20010138; NCT00054379 (obsolete NCT alias)
Record Dates: First submitted 2002-09-06; First posted 2002-09-09 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — epratuzumab

INTERVENTIONS:
Drug: epratuzumab

SUMMARY:
Epratuzumab is currently being studied in combination with rituximab, for the treatment of patients with low-grade NHL who failed previous chemotherapy and have never received rituximab or who received rituximab as a single agent or in combination with chemotherapy as their last treatment and who demonstrated a partial response or complete response for at least 12 months.

ELIGIBILITY:
* Diagnosis of relapsed or refractory low-grade, CD20+, B-cell NHL * Received and failed at least 1 prior regimen of chemotherapy * Rituximab-naive or received prior rituximab in their last treatment (single agent or in combination with chemotherapy) and demonstrated a time to progression of at least 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com